CLINICAL TRIAL: NCT05468034
Title: Exercise in Metastatic Breast Cancer: EMBody
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tarah J Ballinger, MD, Assistant Professor of Clinical Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CTO-IUSCCC-0781
Record Dates: First submitted 2022-07-12; First posted 2022-07-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Indolent Metastatic Breast Cancer
Keywords: breast cancer; indolent metastatic breast cancer; exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): Eligible and consented participants randomized to the exercise arm (EX) will work with an exercise trainer 3x weekly for 16 weeks. Training sessions are 60 min. Schedules are determined by participant and trainer with oversight by the study team, ideally occurring at similar times each day in line with IBC theory. Each training session will be delivered virtually over a HIPAA compliant IU Health Zoom platform. The virtual exercise sessions include 3 parts: cardiovascular exercise, resistance training, and balance or stretching exercise. During sessions, patients will wear provided heart rate monitors with a training goal of moderate intensity, defined as 40-60% of heart rate reserve. Based on the participant's rate of perceived exertion (RPE), heart rate, and individual response during each session, trainers will follow an algorithm designed by the PI and collaborators to progress or regress intensity level. Participant will attend a class on creating and maintaining behavior changes.
  Interventions: Behavioral: Exercise Intervention
- Usual Care (No Intervention): Participants randomized to usual care (UC) will receive care per their treatment team. UC participants are encouraged to exercise but will not be provided components of the intervention. Participants in the UC arm will be given usual care handouts at baseline from the American College of Sports Medicine.

INTERVENTIONS:
Behavioral: Exercise Intervention — Eligible and consented participants randomized to the exercise arm (EX) will work with an exercise trainer 3x weekly for 16 weeks. Training sessions are 60 min. Schedules are determined by participant and trainer with oversight by the study team, ideally occurring at similar times each day in line with IBC theory. Each training session will be delivered virtually over a HIPAA compliant IU Health Zoom platform. The virtual exercise sessions include 3 parts: cardiovascular exercise, resistance training, and balance or stretching exercise. During sessions, patients will wear provided heart rate monitors with a training goal of moderate intensity, defined as 40-60% of heart rate reserve. Based on the participant's rate of perceived exertion (RPE), heart rate, and individual response during each session, trainers will follow an algorithm designed by the PI and collaborators to progress or regress intensity level. Participant will attend a class on creating and maintaining behavior changes.
  Arms: Exercise Intervention

SUMMARY:
The purpose of this study is to study exercise in a novel population with indolent MBC (no progression on current therapy in prior 12 months and not receiving cytotoxic chemotherapy). The study team hypothesizes that delivering virtual, supervised, progressive intensity aerobic and resistance training exercise for 16 weeks in this population will significantly improve 1) cardiorespiratory fitness, functional status, and sarcopenia (low muscle mass), all established predictors of survival, and 2) patient- reported outcomes.

DETAILED DESCRIPTION:
This is a randomized, two arm, single-center study designed to compare the effect of exercise versus usual care control on the clinical parameter of cardiorespiratory fitness, in patients with metastatic breast cancer with indolent disease biology over a 16-week period. This study will be enrolling up to 100 participants. Participants will be randomized 1:1 in blocks of 4 to the exercise intervention or usual care, stratified by frailty yes/no defined by baseline SPPB score ≤ 8 or > 8.

Primary Objective To compare the effect of a 16-week multimodality, virtually delivered exercise intervention on cardiorespiratory fitness measured by a modified Bruce ramp protocol treadmill test to usual care, in patients with indolent metastatic breast cancer.

Secondary Objectives

1. To compare the effect of exercise versus usual care on objective physical function measured by the short physical performance battery (SBBP)
2. To compare the effect of exercise versus usual care on subjective physical functioning measured by PROMIS-29 questionnaire
3. To compare the effect of exercise versus usual care on body composition, measured by visceral adiposity, lean muscle mass, and muscle density on CT scans obtained as standard of care using SliceOmatic software
4. To compare the effect of exercise versus usual care on objective physical activity measured by accelerometer wear
5. To compare the effect of exercise versus usual care on patient reported outcomes, including fatigue (BFI) and health related quality of life (PROMIS-29)
6. To determine the fidelity of the exercise intervention, measured by changes in measures of constructs of habit and intention administered by questionnaire
7. To describe patient uptake and adherence with the intervention, measured by proportion of approached patients who consent to the study, and proportion of assigned training sessions attended by patients randomized to the exercise arm.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Diagnosis of metastatic breast cancer
3. No progression of disease in the 12 months prior to screening per the treating investigator

   1. If participant has changed treatments in the prior 12 months for reasons other than progressive disease, they remain eligible
   2. Participants on no treatment or "no evidence of disease" but still with a diagnosis of metastatic breast cancer are eligible
4. ECOG performance status of 0-2
5. Ability to walk on a treadmill without assistive device.
6. Informed consent and authorization of the release of health information must be obtained according to institutional guidelines
7. Currently not meeting physical activity guidelines (defined as less than 150 minutes of moderate to vigorous exercise per week measured by the IPAQ questionnaire administered during screening)
8. Participants should have a cellular device compatible with iOS 15 or Android operating system 7.

Exclusion Criteria:

1. Receiving cytotoxic chemotherapy at any point in the prior 12 months.

   1. Participants receiving endocrine therapy are eligible.
   2. Participants receiving targeted therapy or antibody therapy are eligible (examples including trastuzumab, pertuzumab, TDM-1, trastuzumab deruxtecan, sacituzumab govetecan, immunotherapy, CDK4/6 inhibitors, olaparib, alpelisib, etc.)
2. Any condition precluding supervised exercise participation. A letter from a physician supporting participation can supersede this eligibility criteria.

   * NYHA class III or IV congestive heart failure
   * Uncontrolled angina
   * Myocardial infarction in the prior 12 months
   * Orthopedic surgery in the previous 3 months or plans for orthopedic surgery during the study period
   * Chronic uncontrolled pulmonary conditions such as uncontrolled asthma (symptoms > 2 days/week) or dyspnea requiring oxygen
   * Symptomatic peripheral vascular disease
   * Or any other comorbidity that would interfere with the ability to complete and comply with the protocol in the opinion of the investigator, including psychological illness
   * History of fragility fracture
3. Active, untreated brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in cardiorespiratory fitness | baseline, 16 weeks
  Measured by minutes on the treadmill

SECONDARY OUTCOMES:
physical performance battery | baseline, 8, and 16 weeks
  total score on short physical performance battery
Mean quality of life, as measured by the Patient-Reported Outcomes Measurement Information System-29 | baseline, 8, and 16 weeks
  Likert-scaled questionnaire, with response scores ranging from 1 to 5. Scores alternate from 1 or 5 being the lowest value.
muscle mass | baseline, and 16 weeks
  measured by mg/kg2 on HU on PET/CT scans
muscle density | baseline, and 16 weeks
  measured by mg/kg2 on HU on CT scans
adipose mass | baseline, and 16 weeks
  measured by mg/kg2 on HU on CT scans
Change in physical activity minutes | baseline to post 16-week intervention
  measured by accelerometer data
Change in steps per day | baseline to post 16-week intervention
  measured by accelerometer data
Mean fatigue score as measured by the Tampa scale for Kinesiophobia (TSK) | baseline, and16-weeks
  17 item Likert scale checklist
Change intention and habits, as measured by the Behavioral Theory Scales | baseline, and 16-weeks
  Likert-scaled questionnaire, measured with a 5-point Likert scale with response options ranging from "strongly disagree" to "strongly agree." Total scores are summed in the range of 40 to 200, with a higher score indicating stronger motivation that could predict exercise behavior.
Uptake of the study | date open to accrual until closed to accrual, up to 2 years
  the proportion of total patients approached, screened, and ultimately completing the baseline assessments
Adherence with the intervention defined | baseline to post 16-week intervention
  the proportion of scheduled sessions attended by participants randomized to the exercise intervention arm
change in patient-reported functional limitations, as measured by a functional limitations scale | baseline, and16-weeks
  mean score of 5 question scale, where participants responses are either scored 0 or 1, with "some difficulty" a 1 and "no difficulty" as a 0.

CONTACTS AND LOCATIONS:
Overall Officials: Tarah Ballinger, MD, Principal Investigator — Indiana University
Locations (6):
- United States (6):
  - Yale Cancer Center, New Haven, Connecticut
  - IU Health West, Avon, Indiana
  - IU Health Joe and Shelly Schwarz Cancer Center, Carmel, Indiana
  - Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Cancilla MA, Nemati D, Halsey D, Shah N, Sherman M, Kelly N, Zhang P, Kassem N, Kaushal N, Shanahan K, Glenn LK, Ligibel JA, Ballinger TJ. Exercise as part of survivorship care in metastatic breast cancer: protocol for the randomized EMBody trial. BMC Cancer. 2024 Sep 12;24(1):1137. doi: 10.1186/s12885-024-12883-6. PMID 39267010